CLINICAL TRIAL: NCT02136810
Title: The Association Between Home Blood Pressures and Clinic Blood Pressures in Patients Presenting for Surgery.
Brief Title: Perioperative Blood Pressures and Chronic Hypertension
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1509016399; K23HL116641 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
Keywords: Hypertension; Perioperative Care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to assess the performance of presurgical clinic blood pressure measurements in predicting home blood pressure readings among surgical patients. It also aims to measure the association between home blood pressures and patient perspectives on blood pressure control.

DETAILED DESCRIPTION:
A convenience sample of presurgical patients seen in a preadmission testing clinic were enrolled and sent home with a home blood pressure monitor that stored up to 50 readings. Participants were asked to return the BP cuff on the day of their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients >= 21 years of age presenting for surgery to a tertiary care preadmission testing clinic.

Exclusion Criteria:

* Inability or unwillingness to independently operate a home blood pressure monitor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory surgical patients >= 21 years of age presenting for preadmission testing to a tertiary care hospital and who demonstrate elevated clinic blood pressures greater than or equal to 130/85mmHg.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schonberger, MD/MHS, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital PreAdmission Testing Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Background] Schonberger RB, Dai F, Brandt CA, Burg MM. Balancing Model Performance and Simplicity to Predict Postoperative Primary Care Blood Pressure Elevation. Anesth Analg. 2015 Sep;121(3):632-641. doi: 10.1213/ANE.0000000000000860. PMID 26214552
- [Background] Schonberger RB, Burg MM, Holt N, Lukens CL, Dai F, Brandt C. The relationship between preoperative and primary care blood pressure among veterans presenting from home for surgery: is there evidence for anesthesiologist-initiated blood pressure referral? Anesth Analg. 2012 Jan;114(1):205-14. doi: 10.1213/ANE.0b013e318239c4c1. Epub 2011 Nov 10. PMID 22075017
- [Background] Schonberger RB. Ideal blood pressure management and our specialty. J Neurosurg Anesthesiol. 2014 Jul;26(3):270-1. doi: 10.1097/ANA.0000000000000012. No abstract available. PMID 24905036

RESULTS

PARTICIPANT FLOW:
Groups:
- Included Participants: A convenience sample of 200 ambulatory patients scheduled for surgery was recruited during their preadmission visit at Yale-New Haven Hospital between November 2015 and December 2016. Inclusion criteria were age ≥21 years and a screening BP ≥ 130/85 mm Hg.
Period: Overall Study
Arm/Group | Included Participants
Started (A convenience sample of 200 participants were enrolled.) | 200
Completed | 200
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Included Participants
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.42 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 185
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 36
  White | 149
  More than one race | 0
  Unknown or Not Reported | 14
SBP [Mean (Standard Deviation); unit: mmHg] | 156.26 (14.11)
DBP [Mean (Standard Deviation); unit: mmHg] | 88.39 (9.81)

OUTCOME MEASURES:

1. Primary Outcome: Performance of Blood Pressure Referral Threshold
Description: The positive predictive value of preadmission testing-measured blood pressure to predict mean home blood pressure >135/85mmHg will be calculated.
Time Frame: Subjects followed for approximately 1 year
Population: Of the 200 participants, 188 returned Home BP Cuffs with valid BP data.
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Included Participants
Number analyzed (Participants) | 188
proportion | .841 [.78 to .89]

2. Secondary Outcome: Patient Perspectives and Beliefs Regarding Blood Pressure Status as They Relate to Actual Home Blood Pressures.
Description: In secondary analyses, the agreement between patients' self-reported blood pressure control (binary outcome) and home blood pressure monitor-determined blood pressure status (binary outcome) will we assessed via Cohen's kappa and raw indices of agreement.
Time Frame: Approximately 60 days
Measure: Number (95% Confidence Interval); unit: Cohen's Kappa coefficient
Arm/Group | Included Participants
Number analyzed (Participants) | 188
Cohen's Kappa coefficient | .158 [.062 to .254]

3. Secondary Outcome: Preidentified Subgroups
Description: The investigators will examine the correlation between blood pressure and heart rate in the subset of patients with hypertension diagnosis.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Patient Perspectives
Description: The possible association of self-reported availability of primary care (5 point LIKERT scale) with home blood pressure monitor-status will be examined by the Mantel-Haenszel Chi-Square Test.
Time Frame: 60 days
Reporting Status: Not Posted

5. Secondary Outcome: Patient Adherence
Description: The possible association of medication adherence (Morisky scale) with home blood pressure monitor-status will be examined by the Mantel-Haenszel Chi-Square Test.
Time Frame: 60 days
Reporting Status: Not Posted

6. Secondary Outcome: Preidentified Subgroup Analysis
Description: The investigators will examine the correlation between blood pressure and heart rate in the subset of patients without hypertension diagnosis.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of enrollment until participant returned for surgery.
Arm/Group | Included Participants
All-Cause Mortality (participants affected / at risk) | 0/200
Serious Adverse Events (participants affected / at risk) | 0/200
Other Adverse Events (participants affected / at risk) | 0/200

LIMITATIONS AND CAVEATS:
94% of participants returned Home BP cuffs with at least one valid reading.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No